CLINICAL TRIAL: NCT03147131
Title: Periprosthetic Bone Mineral Density Changes After Implantation Of A Short Hip Stem Compared To A Straight Stem: Five-Year Results Of A Prospective, Randomized DEXA-Analysis
Brief Title: Periprosthetic Bone Mineral Density Changes After Implantation Of A Short Hip Stem Compared To A Straight Stem
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Ulm (Other)
Responsible Party: Principal Investigator, PD Dr. med Ralf Bieger, PD Dr. med, University Hospital Ulm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D.3067-244/10
Record Dates: First submitted 2016-12-19; First posted 2017-05-10 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis, Hip
Keywords: Total Hip Arthroplasty; Short Stem; DEXA
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fitmore short stem (Active Comparator): Intervention: Total hip arthroplasty with an uncemented femoral short stem, the Fitmore short stem (Zimmer, Warsaw, USA). Furthermore, an uncemented cup (Allofit, Zimmer, Warzaw, USA).
  Device: Fitmore Short Stem
  Interventions: Procedure: Total Hip Arthroplasty
- CLS straight stem (Active Comparator): Intervention: Total hip arthroplasty with an uncemented femoral straight stem, the CLS short stem (Zimmer, Warsaw, USA).Furthermore, an uncemented cup (Allofit, Zimmer, Warzaw, USA).
  Device: CLS Straight Stem
  Interventions: Procedure: Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — Total hip arthroplasty was randomly performed wither either a Fitmore short or a CLS straight stem.

SUMMARY:
The aim of this study is to evaluate periprosthetic bone mineral density (BMD) changes in the proximal femur after implantation of the Fitmore compared to the CLS stem.

DETAILED DESCRIPTION:
After power analysis, 140 consecutive patients were prospectively included in the randomisation protocol receiving either a Fitmore short or a CLS straight stem. The short stem was assigned in 57 (37% females) cases and the straight stem in 83 (38% females) hips. Periprosthetic bone mineral density was measured before surgery, 7 days, 3, 12 and 60 months postoperatively, using dual energy x-ray absorptiometry (DEXA). The results of the first postoperative measurement served as the baseline value. Because of the different length of the two prostheses we used adapted Gruen zones to divide the periprosthetic bone in seven regions of interest (ROI) with equal length in the proximal zones 1,2,6 and 7, only the regions 3 and 5 featured different sizes. Clinical results were recorded using the WOMAC and the Harris hip score (HHS).

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary osteoarthritis of the hip
* written informed consent
* indication for cementless total hip arthroplasty

Exclusion Criteria:

* previous surgery in the same hip
* femoral fracture
* metabolic bone disease
* drugs affecting bone quality
* contralateral THA within the study period
* infectious disease or bony tumor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2010-08-01 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Stem specific stress shielding of a short compared to a straight hip stem | Five years postoperatively
  Periprosthetic Bone Mineral Density changes around a total hip arthroplasty stem

SECONDARY OUTCOMES:
Clinical Outcome after short compared to straight stem THA | Five years postoperatively
  Clinical outcome measured with the Harris Hip Score and the WOMAC

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Bieger, PD Dr., Principal Investigator — University Hospital Ulm - Department of Orthopedic Surgery

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] Freitag T, Hein MA, Wernerus D, Reichel H, Bieger R. Bone remodelling after femoral short stem implantation in total hip arthroplasty: 1-year results from a randomized DEXA study. Arch Orthop Trauma Surg. 2016 Jan;136(1):125-30. doi: 10.1007/s00402-015-2370-z. Epub 2015 Nov 27. PMID 26613788
- [Derived] Meyer JS, Freitag T, Reichel H, Bieger R. Mid-term gender-specific differences in periprosthetic bone remodelling after implantation of a curved bone-preserving hip stem. Orthop Traumatol Surg Res. 2020 Dec;106(8):1495-1500. doi: 10.1016/j.otsr.2020.04.023. Epub 2020 Oct 31. PMID 33132094